CLINICAL TRIAL: NCT00160121
Title: A Phase IV, Open-Label, Multi-Center Trial Evaluating the Efficacy of Fosrenol Compared to Existing Therapy in Adults With End Stage Renal Disease Treated for Hyperphosphatemia
Brief Title: Efficacy and Safety of Fosrenol in Treating Elevated Serum Phosphate Levels in Adults With End Stage Renal Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD405-401
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — lanthanum carbonate

INTERVENTIONS:
Drug: Lanthanum carbonate

SUMMARY:
The purpose of this study is to test how well lanthanum carbonate reduces the pre-dialysis level of serum phosphorus in subjects undergoing dialysis due to end stage renal disease and to determine the patient and physician's satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ESRD who currently require treatment for hyperphosphatemia

Exclusion Criteria:

* Female patient who is pregnant or lactating
* Patient has used any investigational product within 30 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500
Dates: Start 2005-01-10 (Actual); Primary Completion 2005-12-13 (Actual); Study Completion 2005-12-13 (Actual)

PRIMARY OUTCOMES:
Pre-dialysis serum phosphorus levels at 12 weeks | Week 12
Patient satisfaction questionnaire at 12 weeks | Week 12
  7 question patient satisfaction questionnaire for participants to respond to how strongly they agree or disagree with their experience with the medication received in this clinical trial. Question are based on a 4 point ordinal scale of: Strongly Agree, Agree, Disagree, Strongly Disagree.
Physician satisfaction questionnaire at 12 weeks | Week 12
  6 question physician satisfaction questionnaire for physicians to respond to how strongly they agree or disagree with their patient's experience with the medication received in this clinical trial. Question are based on a 4 point ordinal scale of: Strongly Agree, Agree, Disagree, Strongly Disagree.
Patient preference questionnaire at 12 weeks | Week 12
  6 question patient preference questionnaire for participants to respond to whether they preferred the medication they received during this clinical trial or their previous medication.
Physician preference questionnaire at 12 weeks | Week 12
  7 question physician preference questionnaire for physicians to respond to whether they preferred the medication administered during this clinical trial or their patient's previous medication.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

REFERENCES:
- [Result] Wilson RJ, Keith MS, Preston P, Copley JB. The real-world dose-relativity of sevelamer hydrochloride and lanthanum carbonate monotherapy in patients with end-stage renal disease. Adv Ther. 2013 Dec;30(12):1100-10. doi: 10.1007/s12325-013-0077-5. Epub 2013 Dec 5. PMID 24307220
- [Result] Keith MS, Wilson RJ, Preston P, Copley JB. Cost-minimization analysis of lanthanum carbonate versus sevelamer hydrochloride in US patients with end-stage renal disease. Clin Ther. 2014 Sep 1;36(9):1276-86. doi: 10.1016/j.clinthera.2014.06.036. Epub 2014 Jul 26. PMID 25069799
- See also: FDA Recall Information — http://www.fda.gov/opacom/7alerts.html